CLINICAL TRIAL: NCT04259125
Title: Neonatal Seizure Registry: The Role of Inflammation After Neonatal Seizures and Later Development of Epilepsy
Brief Title: Evaluating the Role of Inflammation in Neonatal Epileptogenesis
Acronym: NSR-RISE
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Michigan (Other); Boston Children's Hospital (Other); UCSF Benioff Children's Hospital Oakland (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: K23NS105918 (NIH); K23NS105918 (NIH)
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Neonatal Seizure; Epilepsy; Seizures; Inflammatory Response
Keywords: Neonatal seizure; Inflammation; Cytokine; Micro-RNA; Epilepsy; EEG
MeSH Terms: conditions — Epilepsy; Seizures; Inflammation | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute symptomatic seizures: This is a cohort of 72 participants who will be enrolled into this study from the neonatal intensive care unit (NICU) after being diagnosed with seizures. They will be asked to contribute a blood specimen obtained ideally 48-96 hours (though blood collection allowed 24-120 hours) after seizures are diagnosed, to participate in an optional blood draw at 2-4 months of age, and to complete surveys at 12 & 24 months of age.
  Interventions: Diagnostic Test: Blood draw; Other: Survey
- Control: This is a cohort of 15 participants who will be enrolled into this study from the neonatal intensive care unit (NICU) after having an EEG for possible seizures, but found to have a normal EEG. They will be asked to contribute a blood specimen obtained ideally 48-96 hours (though blood collection allowed 24-120 hours) after birth.
  Interventions: Diagnostic Test: Blood draw

INTERVENTIONS:
Diagnostic Test: Blood draw — Evaluation of plasma inflammatory markers including cytokines and micro-RNA.
Other: Survey — Regarding epilepsy and development.
  Groups: Acute symptomatic seizures

SUMMARY:
The purpose of this study evaluate the relationship between inflammation and epilepsy in neonates with seizures after birth.

DETAILED DESCRIPTION:
Seizures are a common symptom of neurologic dysfunction in the neonatal period, affecting more than 16,000 newborns in the United States per year. Over 25% of neonates with acute symptomatic seizures develop post- neonatal epilepsy (PNE), which is often resistant to medical therapies. There is a critical need to identify those patients most at risk for PNE and understand the mechanisms by which early seizures increase the propensity for recurrent seizures, in hopes of identifying novel therapeutic targets in this population. There is increasing evidence for the role of neuro-inflammation in the development of epilepsy. Levels of cytokines and micro-RNA (miRNA) may serve as markers of disease severity and have been implicated in epileptogenesis in animal models. The purpose of this study is to evaluate plasma cytokine and miRNA levels after neonatal-onset acute symptomatic seizures and determine their association with acute seizure severity and PNE.

ELIGIBILITY:
For participants in the acute symptomatic seizure group:

Inclusion Criteria:

* Neonates <44 weeks corrected age at seizure onset
* Seizures due to acute brain injury
* Parent(s) who are English or Spanish literate (with assistance of interpreter)

Exclusion Criteria:

* Neonates at risk for adverse outcome independent of seizures and underlying brain injury
* Neonates with mild, temporary causes for seizures
* Newborns with neonatal-onset epilepsy syndromes
* Neonates who do not survive the initial hospital admission
* Neonates will not be excluded based on race, ethnicity, gender or gestational age

For participants in the control group:

Inclusion Criteria:

* Neonates that are born > 37 weeks and <44 weeks postmenstrual age at enrollment
* Consultation by the pediatric neurology inpatient service due neonatal paroxysmal events, with normal neurologic examination and ultimate diagnosis of non-epileptic spells on continuous video-EEG (ordered for clinical purposes, not for research) OR consultation for hypoxic ischemic encephalopathy in neonates undergoing therapeutic hypothermia, with early exit from therapy owing to normal neurologic examination, normal continuous video-EEG and uncertain diagnosis of encephalopathy.
* Neonates requiring neurologic consultation for mild hypoxic-ischemic encephalopathy (HIE) undergoing therapeutic hypothermia, with normal examination, cEEG, and neuroimaging upon rewarming.

Ages: 1 Day to 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns who are admitted at one of the participating children's hospitals
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Seizure burden | At study entry
  Investigators will evaluate the seizure burden from the initial diagnostic electroencephalogram (EEG) after birth by determining the average number of seizures per hour.
Percentage of participants diagnosed with epilepsy | 24 months of age
  The investigators will determine the proportion of participants who develop clinical and or electrographic seizures.

SECONDARY OUTCOMES:
Percentage of participants diagnosed with epilepsy | 12 months of age
  The investigators will determine the proportion of participants who develop clinical and or electrographic seizures.
Epilepsy Severity | 12 months of age
  The investigators will administer an investigator-developed questionnaire designed to define the frequency of seizures (monthly, weekly, daily, or greater than daily).
Epilepsy Severity | 24 months of age
  The investigators will administer an investigator-developed questionnaire designed to define the frequency of seizures (monthly, weekly, daily, or greater than daily).
Warner Initial Developmental Evaluation of Adaptive and Functional Skills (WIDEA-FS) | Assessment takes up to 15 minutes and will be conducted at 12 months of age
  The Warner Initial Developmental Evaluation of Adaptive and Functional Skills (WIDEA-FS) will be assessed at 12 months of age. The score ranges from 50 to 200 with higher scores associated with normal development.
Warner Initial Developmental Evaluation of Adaptive and Functional Skills (WIDEA-FS) | Assessment takes up to 15 minutes and will be conducted at 24 months of age
  The Warner Initial Developmental Evaluation of Adaptive and Functional Skills (WIDEA-FS) will be assessed at 24 months of age. The score ranges from 50 to 200 with higher scores associated with normal development.

CONTACTS AND LOCATIONS:
Overall Officials: Adam L Numis, MD, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University of California, San Francisco, San Francisco, California
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Mott Children's Hospital, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Numis AL, Foster-Barber A, Deng X, Rogers EE, Barkovich AJ, Ferriero DM, Glass HC. Early changes in pro-inflammatory cytokine levels in neonates with encephalopathy are associated with remote epilepsy. Pediatr Res. 2019 Nov;86(5):616-621. doi: 10.1038/s41390-019-0473-x. Epub 2019 Jun 24. PMID 31234194